CLINICAL TRIAL: NCT06499259
Title: The Effect of Mandala Coloring Activity on Stress and Anxiety in Mothers With Babies in the Neonatal Intensive Care Unit: A Randomized Controlled Study
Brief Title: The Effect of Mandala Coloring Activity on Stress and Anxiety in Mothers With Babies in NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Prof. Dr., Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/411
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Parents; Psychological Stress
Keywords: Anxiety; Stress; Neonatal Intensive Care Unit; Mandala coloring; Mothers
MeSH Terms: conditions — Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: control group (routine care) and experimental group (mandala painting)
Who Masked: Participant
Masking Description: Stratified and block randomization method will be used in the randomization scheme of the study. In the study, maternal age, number of pregnancies, duration of intensive care unit stay and gestational age variables will be used in the stratification of newborns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Data collection tools will be applied to the mothers in the experimental group and the mandala painting activity will begin. The mandala painting program will consist of a total of 7 mandala painting sessions with 40-minute sessions every day for 7 days. The researcher will accompany the first mandala painting activity. She will answer the participant's questions. The mother will do the remaining 6 mandala coloring sessions alone every day; at the end of the 6 days, the researcher will reapply the data collection tools.
  Interventions: Other: Mandala coloring
- Control group (No Intervention): No application will be made to the mothers in the control group within the scope of the research. Data collection forms will be applied as the first measurement when they are included in the study; at the end of 7 days, the same mothers will fill out the data collection forms again as the last measurement.

INTERVENTIONS:
Other: Mandala coloring — Mandala Pack and Application: The mandala pack is a pack consisting of 7 different patterns suitable for adults and 12 pencils. Mandala patterns will be photocopied by the researcher. Packages will be given to the mothers about mandala coloring and their questions will be answered. The choice of the color of the paint to be used in mandala coloring will be entirely up to the mother. No guidance will be given in this regard.
  Arms: Intervention group

SUMMARY:
The aim of this study was to evaluate the effect of mandala painting activity on stress and anxiety levels in mothers whose babies were hospitalized in the neonatal intensive care unit (NICU).

DETAILED DESCRIPTION:
The health status of the baby and the duration of stay in the intensive care unit cause the mother to experience varying levels of stress and anxiety. It is very important to determine the levels of stress and anxiety in mothers of newborns hospitalized in the Neonatal Intensive Care Unit and to take interventions to reduce it. This study will be conducted to evaluate the effect of mandala coloring activity on stress and anxiety levels in mothers whose babies are hospitalized in the neonatal intensive care unit. It is thought to make an important contribution to the field because it will be a randomized controlled study on the effect of mandala painting activity on stress and anxiety in mothers whose babies are hospitalized in the neonatal intensive care unit.

Type of study: The study was planned as a randomized controlled experimental study.

In the G*Power program, it was determined that it would be sufficient to include 30 participants in the study groups with a 5% alpha margin of error, 0.95 confidence interval, 0.95 effect size and 0.95 power. Considering the randomization list and possible losses, the sample size was increased by 20% and it was decided to include 72 mothers in the study, each group consisting of 36 participants.

Data Collection: Before starting the study, the purpose of the study will be explained to the participant by the researcher and informed consent will be obtained. Data collection tools will be applied to the mothers in the experimental group and the mandala painting activity will begin. The mandala painting program will consist of a total of 7 mandala painting sessions with 40-minute sessions every day for 7 days. The researcher will accompany the first mandala painting activity. She will answer the participant's questions. The mother will do the remaining 6 mandala coloring sessions alone every day; at the end of the 6 days, the researcher will reapply the data collection tools. The mothers in the control group will not receive any treatment within the scope of the study. When they are included in the study, data collection forms will be applied as the first measurement; at the end of 7 days, the same mothers will fill out the data collection forms again as the last measurement. After the completion of the data collection forms, the mothers in the control group will be given a mandala package consisting of 7 applications.

H0: Mandala coloring activity has no effect on stress and anxiety in mothers whose infants are hospitalized in the neonatal intensive care unit.

H1: Mandala coloring activity has a positive effect on stress and anxiety in mothers whose babies are hospitalized in the neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Mothers whose baby has been in the neonatal intensive care unit for at least 3 days and staying in the mother's hotel,
* Having agreed to participate in the research/approved the informed consent form
* No visual or hearing impairment
* Being over 18 years old,
* Being at least literate
* The absence of any problem that would prevent him/her from painting mandala (no problem in his arm or hand that would prevent his movement)
* Must not have a diagnosis of mental illness/anxiety disorder

Exclusion Criteria:

* Mothers with communication and perception problems will not be included in the study.
* Mothers with comprehension and speech problems will not be included in the study.
* Mothers with psychiatric illness and taking medication will not be included in the study.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Before the first mandala painting session (pre-test)
  Visual Analog Scale in the assessment of perceived stress. The use of VAS to assess stress is as discriminative as questionnaires and has construct validity. The VAS used consists of a small dotted ruler with endpoints labeled "no stress" and "maximum stress". Between these two extremes, how much stress is experienced is determined by the VAS. This scale gives a single subjective stress score between 0 and 10.
Visual Analog Scale (VAS) | After the 7th mandala painting session (7 days after the first session) (post-test)
  Visual Analog Scale in the assessment of perceived stress. The use of VAS to assess stress is as discriminative as questionnaires and has construct validity. The VAS used consists of a small dotted ruler with endpoints labeled "no stress" and "maximum stress". Between these two extremes, how much stress is experienced is determined by the VAS. This scale gives a single subjective stress score between 0 and 10.

SECONDARY OUTCOMES:
State Trait Anxiety Inventory (STAI) | Before the first mandala painting session (pre-test)
  The STAI (STAI-State Trait Anxiety Inventory) Scale consist of 20 items each and State Anxiety Scale was used in this study. The State Anxiety Scale has a rating scale consisting of (1) not at all, (2) a little, (3) a lot, (4) completely, according to the degree to which the person feels the current situation. Ten items (items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20) are reverse scored. The cronbach's alpha coefficient of the scale was 0.94 0.96.
State Trait Anxiety Inventory (STAI) | After the 7th mandala painting session (7 days after the first session) (post-test)
  The STAI (STAI-State Trait Anxiety Inventory) Scale consist of 20 items each and State Anxiety Scale was used in this study. The State Anxiety Scale has a rating scale consisting of (1) not at all, (2) a little, (3) a lot, (4) completely, according to the degree to which the person feels the current situation. Ten items (items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20) are reverse scored. The cronbach's alpha coefficient of the scale was 0.94 0.96.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Özdemir, PhD, Study Director — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: September through November of 2025
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data

REFERENCES:
- [Background] Sari Ozturk C, Demir K. The Effect of Mandala Activity and Technology-Based Breastfeeding Program on Breastfeeding Self-Efficacy and Mother-Infant Attachment of Primiparous Women: A Randomized Controlled Study. J Med Syst. 2023 Apr 1;47(1):44. doi: 10.1007/s10916-023-01942-3. PMID 37004692
- [Background] Robinson EM, Baker R, Hossain MM. Randomized Trial Evaluating the Effectiveness of Coloring on Decreasing Anxiety Among Parents in a Pediatric Surgical Waiting Area. J Pediatr Nurs. 2018 Jul-Aug;41:80-83. doi: 10.1016/j.pedn.2018.02.001. Epub 2018 Feb 10. PMID 29439840
- [Background] Ozsavran M, Ayyildiz TK. The effect of mandala art therapy on the comfort and resilience levels of mothers who have children with special needs: A randomized controlled study. Child Care Health Dev. 2023 Nov;49(6):1032-1045. doi: 10.1111/cch.13110. Epub 2023 Mar 16. PMID 36878873